CLINICAL TRIAL: NCT04643119
Title: A Prospective Randomised, Controlled Clinical Trial to Compare the Functional Outcomes of Patients Undergoing Total Knee Replacement Using the Zimmer-Biomet Persona Total Knee System With Cruciate-Retaining or Medial Congruent Bearings
Brief Title: A Comparison of Total Knee Replacement Patients Using the Zimmer-Biomet Persona Total Knee System With Different Inserts
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2020/2866
Record Dates: First submitted 2020-10-25; First posted 2020-11-24 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis, Knee; Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Patients are randomised to 2 different treatment groups by a study team member who will not participate in final data analysis; only their surgeon and the clinical team will be aware of the treatment the patient undergoes. Treatment codes will be used to indicate the patient's treatment assignment in study-related documents, and clinical documents will reference their treatment code as well.
  Radiological, functional and strength assessments will be conducted by non-study clinical staff who will not be aware of the patient's treatment group.
  Analysis will be conducted by a statistician who is uninvolved in the recruitment and data collection process, and only upon completion will the treatment arms will be unblinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cruciate-Retaining Insert (Active Comparator)
  Interventions: Device: Cruciate-Retaining Insert
- Medial-Congruent Insert (Experimental)
  Interventions: Device: Medial Congruent Insert

INTERVENTIONS:
Device: Medial Congruent Insert — The Medial Congruent Bearing (MC Bearing) design was introduced in 2016 for use with the Zimmer-Persona Cruciate-Retaining Femur: the design facilitates greater stability through increased anterior lip height compared to the original Cruciate Retaining Bearing (CR Bearing), allowing for greater anterior constraint and subluxation resistance that aids in full extension and deep flexion. Furthermore, the MC Bearing has been suggested for use in patients presenting with more complicated surgical histories (e.g prior high tibial osteotomies or patellectomies), whereas the original CR Bearing is strictly suggested for use only in patients undergoing knee surgery for the first time, where the posterior cruciate ligament may still be intact.
  Arms: Medial-Congruent Insert
Device: Cruciate-Retaining Insert — The Cruciate-Retaining Bearing (CR Bearing) design was launched together with the use of the Cruciate-Retaining Femoral Components (CR Femur) of the Zimmer-Biomet Persona® Total Knee system. The design not only stabilises the knee through medial conformity and anterior constraint, but also allows for freer and more natural deep flexion through freer movement of the lateral condyle.
  Arms: Cruciate-Retaining Insert

SUMMARY:
As demand for knee joint arthroplasties surge, improving long term patients' satisfaction and implant survivorship has become of utmost importance, as patients seek not only to alleviate their condition, but also return to their usual daily activities and sports. Implant type and design plays an important role in this, with many modern designs seeking to replicate the native knee's kinematics and alignment through mimicry of native knee biomechanics in its femoral components, tibial components, and polyethylene bearing inserts.

The Zimmer-Biomet Persona® Total Knee Cruciate-Retaining Femoral Component (CR Femur), used in conjunction with the kinematic alignment surgical technique, has been shown to produce better functional outcomes and improved patient satisfaction following total knee arthroplasty. More recently, Zimmer-Biomet introduced the Medial Congruent Bearing (MC Bearing) design to be used with the CR Femur; the design facilitates greater stability through increased anterior lip height compared to the original Cruciate Retaining Bearing (CR Bearing), thus allowing for greater anterior constraint and subluxation resistance that aids in activities requiring deeper flexion or full extension. However, the evidence that this will lead to better patient satisfaction and function is scarce, and requires further study to prove that the MC Bearing is a better insert choice to recommend to both surgeons and patients alike.

120 patients from Singapore General Hospital seeking primary total knee replacement surgery will be recruited for this study, and randomised in a 1:1 ratio to receive either the CR Bearing or the MC Bearing alongside the Zimmer-Biomet CR Femur implant. They will be followed up for two years post-operatively, and their outcomes recorded at specific milestones to be analysed for the impact of insert design on knee function, patient satisfaction and quality of life post-surgery.

DETAILED DESCRIPTION:
There has been an increased demand in knee joint arthroplasties, in part due to rising life expectancies and a growing aging population, as well as increased wear and tear in the knees owing to lifestyle factors. As the demand continues to increase annually, improving long term patients' satisfaction and implant survivorship has become of utmost importance, as patients seek not only to alleviate their condition, but also return to their usual, daily activities and sports. Implant design and geometry plays an important role in this, with many modern designs seeking to replicate the native knee's kinematics and alignment through subtle changes in femoral components, tibial components, and polyethylene bearing inserts. The Zimmer-Biomet Persona® Total Knee system tries to replicate the 'feeling' of a native knee through an implant whose design not only stabilises the knee through medial conformity and anterior constraint, but also allows for freer and more natural deep flexion through freer movement of the lateral condyle. The Cruciate-Retaining Femoral Components (CR Femur) of this system, used in conjunction with the kinematic alignment surgical technique, has been shown to produce better functional outcomes and improved patient satisfaction; however, there is a lack of such studies in an Asian population to corroborate these findings.

More recently, Zimmer-Biomet introduced the Medial Congruent Bearing (MC Bearing) design to be used with the CR Femur; the design facilitates greater stability through increased anterior lip height compared to the original Cruciate Retaining Bearing (CR Bearing), thus allowing for greater anterior constraint and subluxation resistance that aids in activities requiring deeper flexion or full extension. Furthermore, the MC Bearing has been suggested for use in patients presenting with more complicated surgical histories (e.g prior high tibial osteotomies or patellectomies), whereas the original CR Bearing is strictly suggested for use only in patients undergoing knee surgery for the first time, where the posterior cruciate ligament may still be intact. This suggests that the MC Bearing may confer better cost-effectiveness, as it may be used in a wider population; combined with its subtle design changes relative to the original bearing design that further enhances the patient's mobility, the MC Bearing may be overall a better insert to recommend to surgeons and patients alike, in the hopes that it would provide the patient a greater degree of mobility, and better satisfaction.

120 patients who are seeking primary TKA surgery in Singapore General Hospital will be recruited to join this study. They will be randomized into two treatment groups in a 1:1 ratio: one group will receive the medial congruent (MC Bearing) polyethylene insert during their surgery, whereas the other group will receive the standard, cruciate-retaining (CR Bearing) design. Randomisation will be carried out by a designated study team member who will not be involved with data collection or data analysis. This team member will also keep the treatment codes in sealed envelopes until the end of the study, where the results can be unblinded, or in extraordinary situations where unblinding of patient is required.

Recruitment is anticipated to take place over twelve months following ethics board approval, beginning in Q1 2021 and completing in Q1 2022. The study is anticipated to complete in two years, with analysis expected to be completed by Q3 2024 following the last participant's last visit at 24 months post-surgery.

All patients in this study will receive routine clinical care pre- and post-operatively from their surgeon for two years; follow-up visits post-surgery will be planned for 1 month, 3 months, 6 months, 12 months and 24 months after surgery. Routine clinical care for patients undergoing TKA surgery include pre-operative and post-operative functional and strength tests at the Orthopaedic Diagnostic Centre, radiological assessments carried out by the Department of Diagnostic Radiology, and consultation visits with the surgeon. Pre-operatively, the patient will also attend a consultation with an anaesthesiologist to confirm their physical fitness for surgery.

Data collected from routine clinical care procedures will be extracted for the purpose of the study. This will include, but is not limited to:

* Preoperative variables: Age at surgery, gender, BMI, side of surgery, American Society of Anesthesiologists (ASA) score, education level, diagnosis, comorbidities including diabetes, heart disease and previous surgical history, preoperative alignment (varus or valgus), range of motion (ankylosed knee), deformity (fixed flexion deformity or recurvatum), preoperative Oxford Knee Score (OKS), Knee Society Function Score (KSFS), Knee Society Knee Score (KSKS), Physical and Mental Component Scores of the 36-Item Health Survey (PCS and MCS respectively), UCLA Activity Score, pain score (using Numerical Pain Rating Scale), and pre-surgery patient expectations and satisfaction(modified rating scale based off the new Knee Society Knee Score)
* Intraoperative variables: polyethylene insert (MC Bearing or CR Bearing)
* Postoperative variables: length of hospital stay, discharge destination, 30 days readmission rate, radiological outcomes such as mechanical axis, coronal femoral component angle, coronal tibial component angle, sagittal femoral component angle, sagittal tibial component angle and change in joint line, postoperative range of motion, residual deformity (fixed flexion deformity or recurvatum), anterioposterior and mediolateral stability of the knee, postoperative OKS, KSFS, KSKS, PCS and MCS, Forgotten Joint Score (FJS), Timed Up And Go (TUG) Test, UCLA Activity Score, complications (deep vein thrombosis/pulmonary embolism, infection, acute myocardial infarction/cerebrovascular accident, postoperative knee stiffness), revision surgery, meeting of expectations and patients' satisfaction

The collated data will be used to analyse if patients in the MC Bearing group experience better functional outcomes and satisfaction. Functional outcome will be scored using the OKS (as the main knee-specific outcome measure), KSFS and KSKS, and TUG score. General health of patients is assessed with the use of the 36-Item Health Survey, modelled after SF-36® (Medical Outcomes Trust, Hanover, New Hampshire, United States), which consists of eight subscales.

In this study, the medical outcome study (MOS) approach was used to derive two higher-order summary scores: PCS and MCS. Meeting of expectations and patients' satisfaction with surgery will be recorded using a scale based off the new Knee Society Knee Score, where patients will be asked 5 questions for expectations, and 5 questions for satisfaction. Responses are scored from 1 to 5 and collated, with higher marks indicating lower satisfaction and met expectations.

During the study's milestone assessments, gait analysis will also be conducted for all patients using GATOR, a non-invasive knee sensor developed by Precision Medical Pte Ltd. The patients will utilise two GATOR units, one for each knee, and carry out four exercises to facilitate data collection: Active Flexion and Extension, Sit-To-Stand-To-Sit, 10-Metre Walk, and Step Up And Step Down. The data collected will be collated and interpreted into a score reflecting the patient's knee health, as well as allow for an objective comparison of the effectiveness of rKA-TKA versus rMA-TKA.

Participants who undergo revision surgery during the course of this study will be analysed for identification of risk factors that could be used in future clinical observations to predict implant survivorship and possibly refine surgical technique.

Statistics will be conducted with an in-house statistician who is not involved in the recruitment or data collection process. All patients' data, inclusive of withdrawn subjects, will be included in the final data analysis as per the intent to treat (ITT) principle. Independent t-tests will be conducted to compare differences in outcomes between the two treatment groups (i.e MC Bearing vs CR Bearing); One-way Repeated Measure ANOVA will be conducted to assess changes in outcomes and patient scores within the group across the timepoints. Non-parametric testing will also be conducted to observe for significant differences in patient outcomes within the groups at each timepoint.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed with, or are experiencing knee osteoarthritis
2. Patients considered fit and appropriate for TKA surgical intervention
3. Patients between 50-80 years of age at time of surgery
4. Patients of Chinese, Malay, or Indian ethnicity (combination of the three groups are accepted)
5. Patient must be capable of giving informed consent and agree to comply with the postoperative review programme
6. Patients who will stay in Singapore for up to two years post-surgery
7. Patients should have sufficient postoperative mobility to attend follow-up clinics and allow for radiographs to be taken
8. Female patients should be post-menopausal, or be willing to take contraceptives/birth control measures throughout study

Exclusion Criteria:

1. Patients not suitable for routine primary TKA e.g. patient has ligament deficiency that requires a constrained prosthesis
2. Patient has bone loss that requires augmentation
3. Patients determined medically unfit for surgical intervention
4. Patients who had prior knee replacement surgery done for the symptomatic limb
5. Patients with impaired musculoskeletal function
6. Patients less than 50 years of age or greater than 80 years of age
7. Patients enrolled on another concurrent clinical trial
8. Patients who are not local residents, or do not intend to stay in Singapore after surgery

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-04-26 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-08-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of Oxford Knee Scores between treatment groups | 2 years
  Differences in total Oxford Knee Scores between the two treatment groups will be compared at 1-month, 3-months, 6-months, 12-months and 24-months post-operatively.
Comparison of Knee Society Rating Scores between treatment groups | 2 years
  Differences in total Knee Society Rating Scores between the two treatment groups will be compared at 1-month, 3-months, 6-months, 12-months and 24-months post-operatively.
Comparison of Forgotten Joint Scores between treatment groups | 2 years
  Differences in total Forgotten Joint- 12 Item Scores between the two treatment groups will be compared at 1-month, 3-months, 6-months, 12-months and 24-months post-operatively.
Comparison of UCLA Activity scores between treatment groups | 2 years
  Differences in total UCLA Activity scores between the two treatment groups will be compared at 1-month, 3-months, 6-months, 12-months and 24-months post-operatively.

SECONDARY OUTCOMES:
Comparison of discharge times between treatment groups | 2 years
  The differences in recovery between patients undergoing total knee arthroplasty with the cruciate-retaining insert, and the patients receiving the same procedure with the medial congruent insert, will be measured through the average Time-To-Discharge from date of surgery between the groups.
Comparison of quality of life between treatment groups | 2 years
  The difference of quality of life will be measured through the overall scores for the eight scales defined in the Short Form Health Survey of 36 Items (SF-36®) assessed at 3-months, 6-months, 12-months and 24-months post-operation, as well as differences in Physical Component Score and Mental Component Score
Comparison of gait in pre-operative and post-operative state | 2 years
  The motion kinematics tracked pre-operatively and post-operatively in the four activities carried out by the patients (Flexion/Extension, Sit-to-Stand-to-Sit, 10-Metre Walk, Step-Up-Step-Down) will be measured using GATOR equipment as provided by Precision Medical Private Limited.

CONTACTS AND LOCATIONS:
Overall Officials: Lincoln Liow, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No